CLINICAL TRIAL: NCT02553135
Title: An Open Label Phase 2 Clinical Trial of Retinal Gene Therapy for Choroideremia Using an Adeno-associated Viral Vector (AAV2) Encoding Rab-escort Protein 1 (REP1)
Brief Title: Choroideremia Gene Therapy Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Byron Lam (Other)
Responsible Party: Sponsor-Investigator, Byron Lam, Professor of Ophthalmology, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150371
Record Dates: First submitted 2015-06-17; First posted 2015-09-17 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Choroideremia
Keywords: choroideremia, gene therapy
MeSH Terms: conditions — Choroideremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Injection of AAV2-REP1 (Experimental): Injection of AAV-REP1, 1.00x10e11 vg, subretinal injection of total volume of 100 μL.
  Interventions: Biological: Injection of AAV2-REP1 (10e11 vg)

INTERVENTIONS:
Biological: Injection of AAV2-REP1 (10e11 vg) — Single Group: single arm study

SUMMARY:
Phase II gene therapy study, involving a total of 6 male patients with choroideremia. The study will be conducted at the Bascom Palmer Eye Institute, University of Miami. Patients will be required to attend a total of 11 study visits over a 24 month period with an additional 3 year follow-up.

DETAILED DESCRIPTION:
This is a Phase II, open label study involving patients with a clinical phenotype of choroideremia and a confirmed CHM genotype. Following consent, patients will be required to attend an initial screening visit (Visit 1). Within 2 weeks of the screening visit patients will undergo a surgical procedure (Visit 2) under general anesthesia which will include a standard vitrectomy, retinal detachment and administration of a subretinal injection of AAV2-REP1 (1x1011 genome particles). Patients will be required to attend a further 9 study visits (Visits 3-11) over a 24 month period for functional, and anatomical assessments as well as monitoring of adverse events. The primary endpoint is the change from baseline in visual acuity in the study eye, compared to control eye. Secondary study endpoints are, change from baseline in autofluorescence evaluation, microperimetry readings and other anatomic and functional outcomes (all in the study eye compared to control eye). Secondary endpoints also include safety assessments to be conducted throughout the study. The fellow eyes of these patients will be utilized as controls in this study and will receive no study treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older
* Male
* Able to give informed consent
* Genetically confirmed diagnosis of choroideremia
* Active disease visible clinically within the macula region
* Best-corrected visual acuity equal to or worse than 20/32 but better than or equal to 20/200 in the study eye.

Exclusion Criteria:

* Female
* Under the age of 18
* History of amblyopia in the study eye
* Men unwilling to use barrier contraception methods
* Relevant grossly asymmetrical disease or other ocular morbidity which might confound use of the fellow eye as a long-term control
* Any other significant ocular and non-ocular disease/disorder or retinal surgery
* Contraindication to use of medications or contrast agents
* Participated in research study involving an investigational product in the past 12 weeks
* Having had gene or cellular therapy at any time prior to this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BYRON LAM, MD, Principal Investigator — UNIVERSITY OF MIAMI, BASCOM PALMER EYE INSTITUTE
Locations (1):
- Bascom Palmer Eye Institute, University of Miami, Miami, Florida, United States

REFERENCES:
- [Derived] Davis JL. The Blunt End: Surgical Challenges of Gene Therapy for Inherited Retinal Diseases. Am J Ophthalmol. 2018 Dec;196:xxv-xxix. doi: 10.1016/j.ajo.2018.08.038. Epub 2018 Sep 5. PMID 30194931

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Injection of AAV2-REP1
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Injection of AAV2-REP1
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Best Corrected Visual Acuity From Baseline
Description: Patients will have an assessment of visual acuity using the Early Treatment of Diabetic Retinopathy Study (ETDRS) vision charts in both eyes. Low Luminance BCVA was measured by placing a 2.0 log unit neutral density filter over the best correction for that eye and having the participant read the normally illuminated ETDRS chart and was reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The study eye was defined as the eye that met inclusion/exclusion criteria with the worst standard BCVA. If the BCVA in both eyes was similar the Patient determines the worse eye be selected as the study eye. A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening.
Time Frame: Baseline, 24 Months
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Injection of AAV2-REP1
Number analyzed (Participants) | 6
Letters | 3.0 (4.0)

2. Secondary Outcome: Change in Retinal Macular Autofluorescence From Baseline
Description: Measured in mm^2 by Fundus Autofluorescence and shows changes in the integrity and metabolism of retinal cells. A negative change from baseline indicates a decrease in size of the retained retina (worsening; disease progression).
Time Frame: 12 and 24 months
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Injection of AAV2-REP1
Number analyzed (Participants) | 6
mm^2
  Baseline to 12 Months | -3.4 (3.6)
  Baseline to 24 Months | 2.8 (2.9)

3. Secondary Outcome: Changes in Microperimetry From Baseline
Description: Microperimetry assessments. A negative change from baseline indicates disease worsening.
Time Frame: Baseline to 24 months
Measure: Mean (Standard Deviation); unit: Average Threshold dB
Arm/Group | Injection of AAV2-REP1
Number analyzed (Participants) | 6
Average Threshold dB | 0.823 (1.789)

4. Secondary Outcome: Number of Participants Who Experience an Adverse Event
Description: Adverse events during treatment and follow-up period
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Injection of AAV2-REP1
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Injection of AAV2-REP1
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Injection of AAV2-REP1 (N=6)
Cataract (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Vitreous Cells (Eye disorders) | 1
Anterior Chamber Cells (Eye disorders) | 1
Extrafoveal macular retinal hole in area of nonfunctioning retina (Eye disorders) | 2
Subretinal fluid (Eye disorders) | 5
Conjunctiva hemorrhage, edema (Eye disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT02553135/Prot_SAP_000.pdf